CLINICAL TRIAL: NCT03052933
Title: Prospective, Multicenter, Open-labeled, Phase I/II Study of the Efficacy and Safety of Copanlisib (BAY 80-6946) and Gemcitabine Combination in Patients With Relapsed/Refractory Peripheral T-cell or NK/T-cell Lymphoma
Brief Title: Copanlisib and Gemcitabine in Relapsed/Refractory PTCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Bayer (Industry); Consortium for Improving Survival of Lymphoma (Other)
Responsible Party: Principal Investigator, Deok-Hwan Yang, Principal investigator, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COPGEM
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Mature T-Cell and NK-Cell Neoplasm
Keywords: copanlisib; gemcitabine; peripheral T-cell lymphoma; extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Extranodal NK-T-Cell | interventions — copanlisib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib/gemcitabine (Experimental)
  Interventions: Drug: Copanlisib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Copanlisib — For phase I study, participants will receive copanlisib (in combination with gemcitabine) IV infusion at a dose of 45 mg or 60 mg on Days 1, 8, and 15 of each 28-day treatment cycle. During phase I study, participants will be treated at the level of 45 mg/dose (level+0), or 60 mg/dose (level+1) of copanlisib. Maximal tolerated dose will be determined by modified 3+3 design including level-1 dose de-escalation.
  For phase II study, copanlisib dose level, determined during phase I study, will be administered on Days 1, 8, and 15.
  Maximum 6 cycles of gemcitabine and copanlisib combination and subsequent copanlisib monotherapy in participants with ≥ SD to copanlisib and gemcitabine until maximum 12 cycles will be given for this study.
Drug: Gemcitabine — For phase I/II study, participants will receive gemcitabine (in combination with copanlisib) IV infusion at fixed dose of 1,000 mg/m2 on Days 1 and 8 of each 28-day treatment cycle until maximum 6 cycles.

SUMMARY:
COPGEM (Copanlisib and Gemcitabine)chemotherapy regimen is proposed as the salvage treatment for relapsed or refractory peripheral T-cell or NK/T-cell lymphomas in this study protocol, which would be expected to be feasible and effective in this group of patients.

Copanlisib (BAY 80-6946), a highly selective and potent class-1 PI3K inhibitor with sub-nanomolar IC50s against PI3Kα and PI3Kδ, has demonstrated activity in relapsed/refractory, aggressive NHLs, suggesting an ORR of 50% for T-cell lymphomas.

Gemcitabine has demonstrated clinical antitumor activity against PTCLs including NK/T-cell lymphomas both as single-agent (ORR 30-50%) and in combination therapy, with limited extramedullary toxicities.

Considering the evidence of activity for both agents against PTCLs, the investigators propose that targeted therapy with copanlisib in combination with gemcitabine will exhibit early elimination of rapidly growing tumor cells and be a rational therapeutic modality for use in relapsed or refractory PTCLs, if the overlapping toxicities can be managed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory PTCL or NK/T-cell lymphomas, excluding primary cutaneous T-cell lymphoma, and Sezary syndrome based on WHO classification,
* Age ≥ 19
* ECOG performance status ≤ 2
* at least one bi-dimensional measurable lesion
* Laboratory values

  * Serum Cr < 1.5 mg/dL or CrCl > 50 mL/min
  * Transaminase (AST/ALT) < 2.5 x ULN (or < 5 x ULN in the presence of lymphoma involvement of the liver)
  * Bilirubin < 1.5 x UNL ( or < 3 x ULN in the presence of lymphoma involvement of the liver or Gilbert syndrome)
  * PT (INR) ≤ 1.5 x ULN and aPTT ≤ 1.5 x ULN
  * Lipase ≤ 1.5 x ULN
  * Hematologic functions: absolute neutrophil count (ANC) ≥ 1,500/µL and platelet count ≥ 75,000/µL, hemoglobin ≥ 8 g/dL
* Left ventricular ejection fraction (LVEF) ≥ the lower limit of normal for the institution
* Women of childbearing potential and men must agree to use adequate contraception when sexually active
* Written informed consent

Exclusion Criteria:

* B-cell NHL, or primary cutaneous T-cell lymphoma and Sezary syndrome
* Patients who had previous history of lymphoma involvement of the CNS.
* History of previous gemcitabine therapy
* Type I or II diabetes mellitus with HbA1c > 8.5% at screening
* History of chronic hepatitis B; subjects positive for HBsAg will be excluded from this study. However, subjects with HBcAb will be eligible if they are negative for HBV DNA quantification
* History of chronic hepatitis C; subjects positive for HCV IgG will be eligible if they are negative for HCV-RNA quantification
* Known history of human immunodeficiency virus (HIV) infection
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* Any other malignancies within the past 3 years except curatively treated basal cell carcinoma of the skin, carcinoma in situ of the uterine cervix, or papillary carcinoma of the thyroid
* Other serious illness or medical conditions

  * Congestive heart failure > NYHA class 2 (Appendix III)
  * Unstable angina or new-onset angina within the last 3 months; Myocardial infarction within 6 months prior to study entry
  * History of significant neurological or psychiatric disorders including dementia or seizure
  * Uncontrolled hypertension despite optimal medical management (per investigator's opinion)
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before start of study treatment
  * Non-healing wound, ulcer, or bone fracture
  * Active uncontrolled infection (viral, bacterial, or fungal infection)
  * Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ grade 3 within 4 weeks of start of study medication
  * Proteinuria estimated by urine protein/creatinine ratio > 3.5 on a random urine sample
  * Concurrent diagnosis of pheochromocytoma
* Other previous or concurrent treatments

  * Ongoing immunosuppressive therapy
  * Radiotherapy or immune-/chemotherapy less than 4 weeks before start of treatment
  * Radioimmunotherapy or autologous transplant less than 3 months before start of treatment
  * Myeloid growth factors within 14 days prior to treatment start
  * Blood or platelet transfusion within 7 days prior to treatment start
  * Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent
  * History of having received an allogeneic bone marrow or organ transplant
  * Major surgical procedure or significant trauma injury within 28 days before start of study medication, open biopsy within 7 days before start of study treatment
  * Anti-arrhythmic therapy (beta-blockers or digoxin are permitted)
  * Use of CYP3A4 inhibitor or inducer
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Concomitant administration of any other experimental drugs under investigation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT), Maximum tolerated dose (MTD) for phase I | 4 weeks
  The recommended dose of the combination of copanlisib and gemcitabine in patients with mature T-cell or NK/T cell neoplasm
Objective response rate for phase II | 1 year
  Primary efficacy data will be maximal change of radiological tumor lesion measurement using CT scan at baseline and every two cycles, with the evaluation of overall response rate, defined as the percentage of patients with a complete response (CR) or a partial response (PR).

SECONDARY OUTCOMES:
adverse events | 2 year
  Toxicity will be graded according to the NCI-CTCAC version 4.0, from the first day of the first cycle of COPGEM chemotherapy to 30 days after the last dose of study drug.
Progression-free survival (PFS) | 2 year
  PFS will be calculated from the start of study drug treatment to the date of disease progression, death, or last follow-up, as appropriate.
Overall survival (OS) | 2 year
  OS will be calculated from the start of study drug treatment to the date of disease death or last follow-up, as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No